CLINICAL TRIAL: NCT06516900
Title: A Comparison of the Effectiveness of OrthoFeet HandsFree Therapeutic Shoes in Reducing Foot Pain and Peak Plantar Pressure
Brief Title: Reducing Foot Pain and Peak Plantar Pressure in Patients With Foot Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Rio Grande Valley (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB 23-0032
Record Dates: First submitted 2024-05-29; First posted 2024-07-24 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Foot Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Own Shoe (No Intervention): Patients wearing their own appropriate shoes
- OrthoFeet shoe (Experimental): Patients wearing OrthoFeet shoes with standard inserts
  Interventions: Device: OrthoFeet HandsFree Therapeutic Shoe

INTERVENTIONS:
Device: OrthoFeet HandsFree Therapeutic Shoe — Patients with foot pain will be recruited for this study and will go for an intervention of wearing OrthoFeet therapeutic shoes for 6 weeks. Each patient will be evaluated and will participate in data collection before and after intervention.
  Arms: OrthoFeet shoe

SUMMARY:
The research project aims to evaluate the effectiveness of OrthoFeet Hands-Free therapeutic shoes and prefabricated inserts in patients with foot pain.

DETAILED DESCRIPTION:
Patients with foot pain frequently have gait dysfunctions resulting in higher mechanical stress and peak plantar pressure in some areas of the foot. Older people with foot pain have impaired balance and reduced walking speed compared to those without foot pain. Higher peak plantar pressure further increases the risk of falls in older populations. By wearing custom-fit devices, such as prefabricated depth shoes, footwear modifications, and orthoses, patients can redistribute pressure by lowering the peak plantar pressure in specific areas. Similarly, these custom-fit devices and shoes may mitigate the level of pain in patients after wearing the shoes for a certain period. Understanding how different orthotics, shoes, and inserts redistribute plantar pressure and lower foot pain is essential to prescribing the proper footwear to foot pain patients. The proposed study will investigate the effectiveness of OrthoFeet Hands-Free therapeutic shoes and prefabricated inserts in patients with foot pain compared to their own shoes. This will be achieved by completing four aims. The first aim will determine the patient shoe wearing compliance, comfort, acceptance, and feasibility of OrthoFeet Hands-Free therapeutic shoes in patients with foot pain. For the second aim, the investigators will determine the effectiveness of reducing foot pain after a 6-weeks intervention of wearing OrthoFeet Hands-Free therapeutic shoes. The third aim will determine the progressive improvements in physical activity, quality of life, and reduction in peak plantar pressure following a 6-weeks intervention period. For the fourth aim, the investigators will compare the effectiveness of reducing plantar pressure between OrthoFeet Hands-Free therapeutic shoes and patients own shoes. The investigators hypothesize that the degree of foot pain mitigates with reduced peak plantar pressure in patients with foot pain after a 6-weeks intervention of wearing OrthoFeet Hands-Free therapeutic shoes greater than occurs when patients continue to wear their own customary shoes. The outcomes from the study will provide a better scenario of how the OrthoFeet shoes and inserts impact the plantar pressure distribution during walking in patients with foot pain. This will further help in future research studies to modify existing designs and guide the development of novel therapeutic treatments for foot pain patients.

ELIGIBILITY:
Inclusion Criteria:

* be able to give written, informed consent
* self-reported foot pain including heel pain, arch or ball of the foot pain, and hallux limitus/rigidus joint pain
* not engaged in any physician prescribed treatment plan
* in-tact protective sensation as determined using Semmes Weinstein monofilament

Exclusion Criteria:

* patients with plantar ulcer
* patients with major foot deformities such as charcot foot, pes cavus
* patients with lower extremity amputation including minor amputation
* foot pain because of nail disorder of keratotic lesions
* patients with unstable conditions such as recent stroke, anticipated changes in medication regime
* acute fractures of the foot
* patients with major cognitive impairment or major depression
* patients with lower extremity decreased protective sensation
* engaged in any treatment of foot pain including icing, oral anti-inflammatories, creams, injections, physical therapy
* swelling

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Foot pain | Baseline, 6 weeks, 12 weeks
  Foot pain will be assessed using the Foot Function Index (FFI) questionnaire. It has three subsections: pain, disability, and activity limitation. The scores for the pain and disability subsections range from 0 to 90 (0 represents best and 90 represents worst), and the score for activity limitation ranges from 0 to 50 (0 represents best and 50 represents worst).
In-shoe Peak Plantar pressure | Baseline, 6 weeks, 12 weeks
  In-shoe peak plantar pressure data will be recorded as patients walk with a pressure-measuring sensor placed inside their shoes. The unit will be Kilopascal (kPa).
Pressure-Time Integral | Baseline, 6 weeks, 12 weeks
  Pressure-Time integral data for different foot regions will be measured as patients walk with a pressure-measuring sensor placed inside their shoes. The unit will be Kilopascal-sec (kPa-s).

SECONDARY OUTCOMES:
Quality of life | Baseline, 6 weeks, 12 weeks
  Medical Outcomes Study 36-item Short Form questionnaires (SF-36) will be used to assess the quality of life. The SF-36 form has four subsections: pain, distance, walking speed, and stair climbing. Each subsection score ranges from 0 to 100 (where 0 is the worst, and 100 is the best health status).
Physical activity | Baseline, 6 weeks, 12 weeks
  Physical activity will be expressed in terms of average steps per day. Patients will wear Actigraph accelerometers for seven consecutive days, and we will record the average steps per day.

CONTACTS AND LOCATIONS:
Locations (1):
- Hafizur Rahman, Harlingen, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified and anonymous dataset will be created for sharing purposes. The dataset will only be shared upon reasonable request and with a written agreement from the recipient. All outcomes, results, and findings will be published in peer-reviewed journals and conference proceedings.
Time Frame: The de-identified and anonymous dataset will only be shared after the study is completed and results are published in peer-reviewed journals and conference proceedings.